CLINICAL TRIAL: NCT06394817
Title: Beijing Disability Risk and Ageing Monitoring Study
Acronym: BEAM
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2022234
Record Dates: First submitted 2024-04-16; First posted 2024-05-01 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-04

CONDITIONS: Age Problem; Disability; Death
Keywords: Disability, Ageing, Cohort
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plan to obtain blood samples from some of the participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total: All subjects
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a community-based prospective cohort study in Beijing, China. The study has been initialized in 2023 and enrolled older residents. This study aims to develop disability risk assessment standards and an early warning model for older adults.

DETAILED DESCRIPTION:
This is a community-based prospective cohort study. Individuals who aged 60 years or older, lived in the communities for more than 1 year, and signed the informed consent form were enrolled in the present study. The study has been initialized in 2023 and aimed to develop an early warning model and a series of disability risk assessment methods for older adults. This work consists of three steps as following. First, we will build a community-based cohort and thus set up a database. Second, an intelligence model for disability risk assessment will be developed using the database. Third, a series of procedures will be established according to the risk assessment model.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Lived in the community for more than 1 year
* Signed the informed consent form

Exclusion Criteria:

* Cannot complete the survey

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community residents aged 60 years or older in China
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2063-05 (Estimated); Study Completion 2063-05 (Estimated)

PRIMARY OUTCOMES:
The prevalence and incidence of functional disability using a population-based survey | An average of 1 to 2 years
  Functional disability was measured by Activities of Daily Living, cognitive function (Mini-Mental State Examination) and movement disorder（Short Physical Performance Battery) collected by questionnaires.The minimum value of the Activities of Daily Living is 0, and the maximum value is 100, the higher the score, the better the outcome.The minimum value of the Mini-Mental State Examination is 0, and the maximum value is 30, the higher the score, the better the outcome.The minimum value of the Short Physical Performance Battery is 0, and the maximum value is 12, the higher the score, the better the outcome.
The prevalence and incidence of mild cognitive impairment using a population-based survey | An average of 1 to 2 years
  Mild cognitive impairment was measured using Mini-Mental State Examination collected by questionnaire.The minimum value of the Mini-Mental State Examination is 0, and the maximum value is 30, the higher the score, the better the outcome.
The prevalence and incidence of dementia using a population-based survey | An average of 1 to 2 years
  Dementia was determined by diagnosis of hospitalization or diagnosis of death or Clinical Dementia Rating scale. The minimum value of the Clinical Dementia Rating is 0, and the maximum value is 3, the higher the score, the worse the outcome.
The conversion rate of normal to mild cognitive impairment | An average of 1 to 2 years
  Percentage of enrolled population that convert from normal to mild cognitive impairment
The conversion rate of mild cognitive impairment to dementia | An average of 1 to 2 years
  Percentage of enrolled population that convert from mild cognitive impairment to dementia
The genetic and environmental factors for mild cognitive impairment and dementia at genomic and expression levels | An average of 1 to 2 years
  Discover risk factors including genetic susceptibility loci (APOE genes and other risk genes) using gene sequencing, cardiovascular risk factors (blood glucose, cholesterol, homocysteine) using laboratory tests, and unhealthy lifestyle using questionnaire.
The biomarkers for normal, mild cognitive impairment, and dementia diagnosis | An average of 1 to 2 years
  Humoral biomarkers are included Aβ42, Aβ40, phosphated tau and total tau in plasma, cerebrospinal fluid, saliva, and urine. Imaging biomarkers are included cerebral volume, glucose metabolism, amyloid and tau deposition of whole brain or hippocampus.
The prevalence and incidence of movement disorder using a population-based survey | An average of 1 to 2 years
  Movement disorder was measured using Short Physical Performance Battery collected by questionnaire.The minimum value of the Short Physical Performance Battery is 0, and the maximum value is 12, the higher the score, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, MD., PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China